CLINICAL TRIAL: NCT02131844
Title: Facilitation of Early Mobilization After Colorectal Surgery: A Randomized Controlled Trial
Brief Title: Early Mobilization After Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Mitacs (Industry)
Responsible Party: Principal Investigator, Dr. Liane S. Feldman, MD, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MUHC Study Code 13-329-SDR; Mitacs Elevate Fellowship (Other Grant/Funding Number: IT02887)
Record Dates: First submitted 2014-03-28; First posted 2014-05-06 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Colonic Diseases; Rectal Diseases
Keywords: colorectal surgery; postoperative recovery; early mobilization
MeSH Terms: conditions — Colonic Diseases; Rectal Diseases | interventions — Early Ambulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Facilitated early mobilization (Experimental): Early mobilization facilitated by a dedicated health professional
  Interventions: Other: Facilitated early mobilization
- Usual care (Active Comparator): Instructions about early mobilization covered in a preoperative education session
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Facilitated early mobilization — Participants randomized to this group, in addition the preoperative education (usual care), will have early mobilization facilitated by a trained health professional. This health professional will: (1) visit the participant on the day of surgery to reinforce mobilization goals and assist with transfer to a chair and (2) visit the participant three times per day starting from POD 1 to reinforce mobilization goals and walk with the participant (at least the length of the hallway). Targeted walking distances will increase according to the participant's tolerance. This intervention will be undertaken until POD 3 or hospital discharge, whichever comes first.
  Other Names: Early ambulation
  Arms: Facilitated early mobilization
Other: Usual care — Participants randomized to this group will receive instructions about postoperative mobilization in a preoperative education session and will receive a booklet describing mobilization goals for each POD (sit in a chair for 2 hours on the day of surgery, stay out of bed for at least 6 hours/day from POD 1 until hospital discharge)
  Other Names: Preoperative education
  Arms: Usual care

SUMMARY:
Early mobilization (i.e. initiation of out of bed activities from the day of surgery) is considered an important component of postoperative care after colorectal surgery. Having a health professional dedicated to facilitate early mobilization has the potential to enhance postoperative recovery by preventing the negative effects of prolonged bed rest (e.g. increased risk for complications, muscle loss, deconditioning and functional decline); however, the need to implement this resource-intensive approach is not evidence based. This study aims to contribute evidence about the role of facilitated early mobilization as a strategy to enhance recovery after colorectal surgery.

DETAILED DESCRIPTION:
The primary research question of this study is: to what extent does postoperative facilitation of early mobilization impact on recovery of functional walking capacity at 4 weeks after surgery in comparison to standard care (preoperative education).

The hypothesis is that, by 4 weeks after surgery, facilitated early mobilization will result in a greater proportion of participants returning to preoperative levels of functional walking, as measured by the six-minute walk test (6MWT).

ELIGIBILITY:
Inclusion Criteria:

* Adult people (>18 years)
* Colonic or rectal diseases (i.e. cancer, inflammatory bowel disease, diverticulitis) planned for surgical resection

Exclusion Criteria:

* Metastatic disease
* Medical conditions that preclude postoperative mobilization (e.g. neurological or musculoskeletal diseases)
* Inability to understand English or French
* Admission to intensive care immediately after the surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-08; Primary Completion 2015-07 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Functional walking capacity (six-minute walk test) | before surgery; 4 weeks after surgery
  The outcome of interest will be the proportion of participants returning to preoperative levels of functional walking capacity at 4 weeks after surgery (within an estimated measurement error of 20 meters)

SECONDARY OUTCOMES:
Time out of bed (sitting and standing) | postoperative day (POD) 0, 1, 2 and 3
  Measured by an activity monitor (Actigraph) worn over the participants' hip
Time to readiness for discharge | duration of hospital stay (expected average of 3 days after surgery)
  Time to achieve standardized hospital discharge criteria (tolerance of oral intake, recovery of lower gastrointestinal function, adequate pain control on oral analgesia, ability to mobilize and self care and no evidence of complications or untreated medical problems).
Time to recovery of gastrointestinal motility | Expected average of 2 days after surgery
  Time to achieve criteria for recovery of gastrointestinal transit (tolerance of solid diet and bowel movement)
Postoperative fatigue (Multidimensional Fatigue Inventory) | before surgery; POD 1, 2 and 3; 2 weeks after surgery; 4 weeks after surgery.
Self-reported physical activity status (Duke Activity Status Index) | before surgery; 2 weeks after surgery; 4 weeks after surgery
Mobility (Life-Space Mobility Assessment) | before surgery; 4 weeks after surgery
Condition-specific health-related quality of life (Abdominal Surgery Impact Scale) | before surgery; POD 1, 2 and 3; 2 weeks after surgery; 4 weeks after surgery
Generic heath-related quality of life (RAND-36) | before surgery; 4 weeks after surgery
Postoperative complications | up to 4 weeks after surgery
  Classified according to Clavien-Dindo Index and converted into a continuous scale using the Comprehensive Complication Index
Pulmonary function (spirometry) | before surgery; POD 1, 2 and 3; 4 weeks after surgery
  Forced vital capacity (FVC), forced expiratory volume in one second (FEV1) and cough expiratory flow (CEF) will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Liane S Feldman, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Julio F Fiore Junior, PhD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Nancy Mayo, PhD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Franco Carli, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Balvardi S, Pecorelli N, Castelino T, Niculiseanu P, Alhashemi M, Liberman AS, Charlebois P, Stein B, Carli F, Mayo NE, Feldman LS, Fiore JF Jr. Impact of Facilitation of Early Mobilization on Postoperative Pulmonary Outcomes After Colorectal Surgery: A Randomized Controlled Trial. Ann Surg. 2021 May 1;273(5):868-875. doi: 10.1097/SLA.0000000000003919. PMID 32324693
- [Derived] Fiore JF Jr, Castelino T, Pecorelli N, Niculiseanu P, Balvardi S, Hershorn O, Liberman S, Charlebois P, Stein B, Carli F, Mayo NE, Feldman LS. Ensuring Early Mobilization Within an Enhanced Recovery Program for Colorectal Surgery: A Randomized Controlled Trial. Ann Surg. 2017 Aug;266(2):223-231. doi: 10.1097/SLA.0000000000002114. PMID 27997472